CLINICAL TRIAL: NCT01610141
Title: Applying Pharmacogenetics to Warfarin Dosing in Chinese Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Tong Yin, Institute of Geriatric Cardiology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSFC-30971259
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Pulmonary Embolism; Heart Valve Disease
Keywords: warfarin metabolism; pharmacogenetics; CYP2C9; genotyping; VKORC1; CYP4F2; anticoagulation; atrial fibrillation; deep vein thrombosis; pulmonary embolism; Artificial Heart Valve
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism; Heart Valve Diseases; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genotype-guided warfarin dosing (Experimental): A pharmacogenetic dosing algorithm including clinical factors and genotype information (VKORC1, CYP2C9 and CYP4F2) will be used to determine warfarin doses.
  Interventions: Other: Genotype-guided warfarin dosing
- Non-genotype guided warfarin dosing (Active Comparator): A fixed warfarin dose of 3 mg/day was given to the patients for at least 3 days. Following doses were adjusted according to the INR measurement.
  Interventions: Other: Non-genotype guided warfarin dosing

INTERVENTIONS:
Other: Genotype-guided warfarin dosing — Applying a Pharmacogenetic-guided warfarin dosing algorithm derived from Chinese to determine the daily maintenance dose of warfarin, based on clinical factors (age, sex, body surface area, etc.), and VKORC1, CYP2C9 and CYP4F2 genotypes, to individualize the dosing of warfarin.
  Arms: Genotype-guided warfarin dosing
Other: Non-genotype guided warfarin dosing — A Empiric fixed warfarin dose of 3 mg/day was given to the patients for at least 3 days. Following doses were adjusted according to the INR measurement.
  Arms: Non-genotype guided warfarin dosing

SUMMARY:
The purpose of this study is to determine whether pharmacogenetic guided dosing of warfarin is promising for the improvement of efficiency, therapeutic efficacy, and, especially, safety of warfarin therapy than a dosing regimen without the pharmacogenetic information in Chinese patients initiated on warfarin anticoagulation.

DETAILED DESCRIPTION:
Warfarin is the most widely used oral anticoagulation drug for preventing and treating thromboembolic events, but there is greater than 10-fold interindividual variability in the dose required to attain a therapeutic response. In 2007, the US Food and Drug Administration updated the label of warfarin, recommending consideration of pharmacogenetic information which has been confirmed to contribute significantly to the variability in warfarin dose requirements. Thereafter, multiple pharmacogenetic dosing algorithms were constructed to predict warfarin dose by integrating clinical and genetic factors. Taken together, approximately between one-third and one- half of the variability in warfarin dose could be explained by the proposed algorithms. However, the potential benefit of these dosing algorithms in terms of their safety and clinical utility has not been adequately investigated in randomised settings in Chinese patients.

Study objectives:

1. To apply routine pharmacogenetic (PG)-guided dosing of warfarin in clinical practice in Chinese patients.
2. To compare the percentage out-of-range (%OOR) International Normalized Ratios (INRs) during the first 3 month of warfarin therapy using PG-guided dosing with historical standard (STD), empiric dosed controls.
3. To compare the cost effectiveness, number of thromboembolic and bleeding events, time within therapeutic INR range, time to reach stable dose and number of supratherapeutic INR peaks during the first 3 month of warfarin therapy using PG-guided dosing with historical standard (STD), empiric dosed controls.

Study design:

This is a prospective, randomized study of Chinese patients who are to initiate chronic warfarin anticoagulation for specific, qualifying clinical reasons (i.e., atrial fibrillation, Deep vein thrombosis/pulmonary embolism, or Prosthetic valve replacement). Qualifying patients will be consented and randomized to an individualized, pharmacogenetic guided warfarin-dosing regimen (PG group) or to standard care (without knowledge of genotype)(STD group). All patients will receive a baseline INR. For patients in PG group, a maintenance dose for each patient will be predicted by the pharmacogenetic algorithm derived previously in Chinese. A maintenance dose of 3 mg/day will designed to each patients in STD group. The starting dose of warfarin that is twice the assigned daily maintenance dose will be prescribed on the first and second days, and then the dose will revert to the assigned maintenance dose.

Study duration:

Each patient will participate for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Patients initiated on warfarin for venous thromboembolism, pulmonary embolism, atrial fibrillation or heart valve replacement that require long- term oral anticoagulation with target INR ranged 1.5-3.0 for at least 3 months
* Ability to attend scheduled visits
* Signed informed consent

Exclusion Criteria:

* Non-eligible subject
* Pregnant,lactating or of child-bearing potential women
* Patients with severe co-morbidities (e.g., renal insufficiency/creatinine > 2.5 mg/dL,hepatic insufficiency, active malignancy, terminal disease)
* Known genotype CYP2C9 or VKORC1 at start of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
A comparison between the pharmacogenetic and standard arms of the per-patient percentage of out-of-range INRs (<1.5, >3). | 3 months

SECONDARY OUTCOMES:
Time to the first supratherapeutic INR | 3 months
The proportion of time within the therapeutic INR range | 3 months
The proportion of patients reaching therapeutic INR on days 5 and 8 | 3 months
The total number of INR measurements and number of dose adjustments made | 3 months
Proportion of INRs > 4 | 3 months
Major bleeding events | 3 months
Minor bleeding events | 3 months
Thromboembolic complications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tong Yin, Dr., Principal Investigator — Institute of Geriatric Cardiology, General Hospital of People's Liberation Army, Beijing China
Locations (1):
- Institute of geriatric Cardiology, General Hospital of People's Liberation Army, Beijing, China

REFERENCES:
- [Background] Liu Y, Yang J, Xu Q, Xu B, Gao L, Zhang Y, Zhang Y, Wang H, Lu C, Zhao Y, Yin T. Comparative performance of warfarin pharmacogenetic algorithms in Chinese patients. Thromb Res. 2012 Sep;130(3):435-40. doi: 10.1016/j.thromres.2012.02.003. Epub 2012 Feb 27. PMID 22374335